CLINICAL TRIAL: NCT04643106
Title: A Multi-center, Randomized, Investigator-initiated Trial to Evaluate the Efficacy of PRreservation of ovArian Function, Hemostasis, and sAfety of a Hemostatic Agent Versus Suturing During Laparoscopic Ovarian Cystectomy for Endometrioma
Brief Title: Comparison of Hemostatic Agent to Suture in Terms of Hemostatic Function and Preservation of Ovarian Function
Acronym: PRAHA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-059-1147
Record Dates: First submitted 2020-11-01; First posted 2020-11-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Benign Ovarian Cyst
Keywords: endometriosis; endometrioma; ovarian cystectomy; ovarian function; ovarian reserve; hemostatic agent; suture
MeSH Terms: conditions — Endometriosis | interventions — Hemostasis; Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemostatic agent group (Experimental): During laparoscopic ovarian cystectomy, bleeding will be controlled by using a hemostatic agent (EVICEL® Fibrin Sealant, Ethicon, USA), which consist of thrombin and coagulating proteins, mainly fibrinogen and fibronectin. If hemostasis is not fulfilled enough by using it, a additional intervention such as electrocoagulation with bipolar forceps and barbed suture is required to stop bleeding.
  Interventions: Procedure: Hemostatic agent (EVICEL®) application during laparoscopic ovarian cystectomy
- Suturing group (Active Comparator): During operation, barbed suture will be applied to the inner surface of ovarian parenchyme where ovarian endometriosis was attached. In this group, if bleeding is continued after suturing, additional electrocoagulation with bipolar forceps will be conducted.
  Interventions: Procedure: suturing with barbed sutures during laparoscopic ovarian cystectomy

INTERVENTIONS:
Procedure: Hemostatic agent (EVICEL®) application during laparoscopic ovarian cystectomy — During laparoscopic ovarian cystectomy, bleeding will be controlled by using a hemostatic agent (EVICEL®)
  Arms: Hemostatic agent group
Procedure: suturing with barbed sutures during laparoscopic ovarian cystectomy — During laparoscopic ovarian cystectomy, suturing of ovarian inner surface will be conducted to stop bleeding
  Arms: Suturing group

SUMMARY:
This study aims to evaluate the efficacy of preservation of ovarian function, hemostasis, and safety of a hemostatic agent versus suturing during laparoscopic ovarian cystectomy for ovarian endometriosis.

DETAILED DESCRIPTION:
In women with endometrioma who plan to undergo laparoscopic ovarian cystectomy, surgical technique can influence postoperative ovarian function because of removal of normal ovarian tissue with ovarian cyst and damage to ovarian tissue during bleeding control after stripping of endometrioma. This study is designed to compare hemostatic sealant to suturing in terms of hemostatic function, safety and preservation of ovarian function.

Ovarian function of all patients will be evaluated on pre op, post op 12 weeks, post op 48 weeks by measuring AMH and ovarian volume. And Hemostatic function will be evaluated by measuring serum hemoglobin, blood loss during operation, etc.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Age: 19-45 year-old women
* American Society of Anesthesiologists Physical Status classification 1 or 2
* Plan of laparoscopic ovarian cystectomy for unilateral or bilateral ovarian endometriosis diagnosed by ultrasonography
* Regular menstruation every 21-45 days

Exclusion Criteria:

* No 'ovarian' endometriosis
* Suspicious disease of ovarian malignancy
* Age: 18 and younger, 46 and older
* Pregnancy or breastfeeding.
* Lower than 0.05 ng/ml of serum Anti-mullerian hormone level
* Hormonal therapy within recent 3 months
* Considered as inappropriate by the researcher's judgment.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ovarian function preservation 12 weeks after surgery | 12 weeks after surgery
  Reduction rate of AMH level in serum 12 weeks after surgery

SECONDARY OUTCOMES:
Ovarian function preservation 48 weeks after surgery | 48 weeks after surgery
  Reduction rate of AMH level in serum 48 weeks after surgery
The time required to finish hemostasis | during operation
  Stop-watch will be operated right after finishing stripping endometrioma. It will be evaluated how long the time have been spent for bleeding control
the success rate of hemostasis within 10 minutes | during operation
  Stop-watch will be operated right after finishing stripping endometrioma. It will be evaluated whether hemostasis is finished within 10 minutes
Blood loss during operation | during operation
  The volume of blood loss will be estimated by using simple visual assessment technique referring to gauze count and irrigation bottle
Hemoglobin | post-op 2 days, 12 weeks and 48 weeks
  Change of serum hemoglobin from baseline
Transfusion during admission | post-op 2 days
  whether patients are transfused during admission period
Adverse events associated with operation, bleeding or transfusion | post-op 2 days
  any adverse events during admission period
Hospitalization period | within post-op 2 weeks
  days from admission day to discharge day
Operation running time | during operation
  time from anesthesia start to delivery of patient to recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Hee seung Kim, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim H, Park SJ, Paik H, Mun J, Lee EJ, Lee S, Lim W, Song G, Shim SH, Lee CH, Yim GW, Kim HS; PRAHA Study Group. Preservation of the ovarian reserve and hemostasis during laparoscopic ovarian cystectomy by a hemostatic agent versus suturing for patients with ovarian endometriosis: study protocol for randomized controlled, non-inferiority trial (PRAHA-2 trial). Trials. 2021 Jul 21;22(1):473. doi: 10.1186/s13063-021-05431-1. PMID 34289889